CLINICAL TRIAL: NCT05259163
Title: An Evaluation of the LFR-260 Against a Traditional Phoropter in Visual Acuity Testing
Brief Title: LFR-260 vs Traditional Phoropter in Visual Acuity Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evolution Optiks Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: LFR-260-2021
Record Dates: First submitted 2022-02-09; First posted 2022-02-28 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Visual Acuity; Astigmatism; Anisometropia
Keywords: Ocular
MeSH Terms: conditions — Astigmatism; Anisometropia

STUDY DESIGN:
Intervention Model Description: The investigational product was compared to the traditional phoropter. Subjects were randomized to the order of testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Group 1: LFR-260 first, then traditional phoropter (Experimental): The LFR-260 was administered first in this group, followed by the traditional phoropter. The LFR-260 is a portable digital refractor which allows for determination of refractive error as well as for fully remote refractions during eye exams. The traditional phoropter is intended to be used for distance vision testing in any environment.
  Interventions: Device: LFR-260 portable phoropter; Device: Traditional phoropter (SOC)
- Group II: Traditional Phoropter first, then LFR-260 (Active Comparator): The traditional phoropter was administered first in this group, followed by the traditional phoropter. The traditional phoropter is intended to be used for distance vision testing in any environment. The LFR-260 is a portable digital refractor which allows for determination of refractive error as well as for fully remote refractions during eye exams.
  Interventions: Device: LFR-260 portable phoropter; Device: Traditional phoropter (SOC)

INTERVENTIONS:
Device: LFR-260 portable phoropter — Portable unit to evaluate visual refractive state of the patient
Device: Traditional phoropter (SOC) — Standard unit for evaluating visual refractive state of the patient

SUMMARY:
The purpose of this study is to establish if LFR-260 (investigational device) is not inferior in effectiveness to a traditional phoropter (control device) when applied in visual acuity test in subjects undergoing a full routine eye examination. LFR-260 proposes to provide information of the visual capabilities of the patient. The test will be provided and supervised by a qualified eye care provider. The informed consent, screening, randomization (into the order of visual test device used), (visual) device testing (to include precision testing, remote and offsite testing) will all occur at a single visit.

ELIGIBILITY:
Inclusion Criteria:

1. The participant or legal guardian is willing and able to understand, sign and date the Ethics committee approved study specific Informed Consent Form.
2. The participant is a male or female between the ages of 12 and 65 (inclusive).
3. The participant has no more than mild to moderate far-sightedness, near-sightedness, astigmatism or anisometropia.
4. The participant is free of ocular and systemic abnormalities that might affect visual functions.

Exclusion Criteria:

1. The participant has diabetes mellitus (Type 1 or 2).
2. The participant has an autoimmune condition.
3. The participant is pregnant (self-reported).
4. The participant has an active corneal or conjunctival infection.
5. The participant has an active corneal, conjunctival, or intraocular inflammation (i.e. - uveitis).
6. The participant has diabetic retinopathy.
7. The participant has glaucoma or ocular hypertension.
8. The participant has macular degeneration.
9. The participant has had a previous ocular surgery.
10. The participant has ocular and systemic diseases or abnormalities that might affect visual functions.
11. The participant has a history of amblyopia, strabismus, or any other binocular vision abnormality.
12. The participant has a history of AMD (age macular degeneration).
13. The participant is a prisoner, a transient or has been treated for alcohol and/or drug abuse in an inpatient substance abuse program within 6 months prior to proposed study enrolment.
14. The participant will not be able to complete questionnaires.
15. The participant is currently in an investigational study for a similar purpose.
16. The participant, in the judgment of the Investigator, may be inappropriate for the intended study procedures.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MCPHS, Worcester, Massachusetts
  - Gold Coast Optometric Vision, Oyster Bay, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- LFR-260 First, Then Traditional Phoropter: The LFR-260 was administered first in this group, followed by the traditional phoropter. The LFR-260 is a portable digital refractor which allows for determination of refractive error as well as for fully remote refractions during eye exams.
  LFR-260 portable phoropter: Portable unit to evaluate visual refractive state of the patient
- Traditional Phoropter First, Then LFR-260: The traditional phoropter was administered first in this group, followed by the LFR-260. The traditional phoropter is intended to be used for distance vision testing in any environment. The traditional phoropter is an application-controlled instrument providing the same subjective refraction capabilities for distance vision testing as the standard of care eye examination including sphere, cylinder, and axis. Traditional phoropter (Standard of Care): Standard unit for evaluating visual refractive state of the patient
Period: Initial Testing - 1st Intervention
Arm/Group | LFR-260 First, Then Traditional Phoropter | Traditional Phoropter First, Then LFR-260
Started | 56 | 56
Completed | 55 | 56
Not Completed | 1 | 0
Not completed — Investigator needed to continue adding cylinder beyond testing limit for the device. | 1 | 0
Period: 1 Hour (+/- 30 Min) - 2nd Intervention
Arm/Group | LFR-260 First, Then Traditional Phoropter | Traditional Phoropter First, Then LFR-260
Started | 55 | 56
Completed | 55 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group I: LFR-260 First, Then Traditional Phoropter: The LFR-260 was administered first in this group, followed by the traditional phoropter.
- Group II: Traditional Phoropter First, Then LFR-260: The traditional phoropter was administered first in this group, followed by the LFR-260.
- Total: Total of all reporting groups
Arm/Group | Group I: LFR-260 First, Then Traditional Phoropter | Group II: Traditional Phoropter First, Then LFR-260 | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Customized [Count of Participants; unit: Participants]
  Age Category: <=21 years | 16 | 10 | 26
  Age Category: >21 years | 39 | 46 | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 22
  Not Hispanic or Latino | 42 | 47 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 10 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 34 | 39 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 55 | 56 | 111

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of LFR260 on Visual Acuity Test
Description: Agreement of LFR-260 (investigational device) to traditional phoropter (comparator device) when applied in visual acuity test (eye chart test) in subjects undergoing a full routine eye examination. Agreement will be determined by demonstrating that the LFR-260 is within 0.5D (+/-) in measuring sphere and cylinder results and within 10 degrees for axis results among subjects with low astigmatism and within 5 degrees among subjects with moderate to high astigmatism from the traditional phoropter.
Time Frame: Day 0
Population: The total number of eyes analyzed was 222 for 111 study participants.
Measure: Number; unit: percentage meeting criteria
Units Other Than Participants: eyes
Groups:
- Group I: The LFR-260 was administered first in this group, followed by the traditional phoropter.
- Group II: The traditional phoropter was administered first in this group, followed by the LFR-260.
Arm/Group | Group I | Group II
Number analyzed (Participants) | 55 | 56
Number analyzed (eyes) | 110 | 112
percentage meeting criteria | 76.6 | 76.6

2. Primary Outcome: Precision of LFR260 in Repeated Testing
Description: Precision testing will also be conducted to confirm repeatability and reproducibility of the LFR-260.
Time Frame: Day 0
Measure: Number (90% Confidence Interval); unit: percentage meeting criteria
Units Other Than Participants: eyes
Arm/Group | Group I | Group II
Number analyzed (Participants) | 55 | 56
Number analyzed (eyes) | 110 | 112
percentage meeting criteria | 93.8 [89.3 to 96.7] | 93.8 [89.3 to 96.7]

3. Secondary Outcome: Patient Satisfaction Survey
Description: 4-question survey (1=worst; 5=best) given to patients to determine satisfaction with LFR-260 device Quad view.
  Q1: Was the LFR-260 device Quad view comfortable to use for your eye exam? (1=very uncomfortable - 5=very comfortable) Q2: Did the LFR-260 Quad view feel the same as the traditional phoropter when taking your eye exam? (1=LFR-260 definitely more uncomfortable - 5=LFR-260 definitely more comfortable) Q3: Did you prefer to read the eye chart using the LFR-260 device Quad view or traditional phoropter? (1=definitely prefer phoropter - 5=definitely prefer LFR-260) Q4: If taking an eye exam in the future, would you prefer your doctor use the LFR-260 Quad view or traditional phoropter? (1=definitely prefer phoropter - 5=definitely prefer LFR-260)
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I | Group II
Number analyzed (Participants) | 55 | 56
score on a scale
  Question 1 | 3.7 (.93) | 3.6 (1.05)
  Question 2 | 2.5 (1.35) | 2.5 (1.16)
  Question 3 | 2.1 (1.51) | 2.1 (1.41)
  Question 4 | 2.3 (1.31) | 2.3 (1.33)

4. Secondary Outcome: Provider Satisfaction Survey
Description: 4-question survey (1=worst; 5=best) given to eye care provider to determine satisfaction with LFR-260 related to usability, convenience.
  Q1: LFR-260 device performed as expected according to the Instructions for Use (IFU)? (1=definitely did not - 5=definitely) Q2: LFR-260 device was easy to use? (1=very difficult to use - 5=very easy to use) Q3: LFR-260 device was intuitive to operate? (1=definitely counterintuitive - 5=very intuitive) Q4: LFR-260 was more or less convenient to use than the phoropter? (1=definitely less convenient- 5=definitely more convenient)
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I | Group II
Number analyzed (Participants) | 55 | 56
score on a scale
  Question 1 | 4.4 (1.03) | 4.4 (1.12)
  Question 2 | 3.8 (1.20) | 3.7 (1.2)
  Question 3 | 3.1 (1.10) | 3.0 (1.04)
  Question 4 | 2.3 (.75) | 2.2 (.78)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the study period for each patient, which included a single visit where all study data was collected, up to 4 hours.
Groups:
- LFR-260: The LFR-260 is a portable digital refractor which allows for determination of refractive error as well as for fully remote refractions during eye exams.
  LFR-260 portable phoropter: Portable unit to evaluate visual refractive state of the patient
- Traditional Phoropter: The traditional phoropter is intended to be used for distance vision testing in any environment. The traditional phoropter is an application-controlled instrument providing the same subjective refraction capabilities for distance vision testing as the standard of care eye examination including sphere, cylinder, and axis.
  Traditional phoropter (Standard of Care): Standard unit for evaluating visual refractive state of the patient
Arm/Group | LFR-260 | Traditional Phoropter
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT05259163/Prot_SAP_001.pdf